CLINICAL TRIAL: NCT05332301
Title: Exploring Sex Differences in the Acute Postprandial Metabolic Response to a High-fat Mixed Macronutrient Meal Challenge in Healthy Young Humans
Brief Title: Sex Differences in Metabolism Following a High-fat Meal
Acronym: HFM
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Kirsten Bell (Other)
Collaborators: McMaster University (Other)
Responsible Party: Sponsor-Investigator, Kirsten Bell, Assistant Professor, McMaster University
Organization: McMaster University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 14714
Record Dates: First submitted 2022-04-08; First posted 2022-04-18 (Actual); Last update posted 2025-08-19 (Actual); Status verified 2025-08

CONDITIONS: Healthy Nutrition
Keywords: glucose metabolism; lipid metabolism; substrate oxidation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- High-fat test meal (Experimental): All participants will consume a high-fat breakfast after an overnight fast. This meal will consist of a flour tortilla, eggs, bacon, cheddar cheese, mayonnaise, and hashbrowns. After the initial blood sample (0 min) is drawn during Visit 2, we will ask participants to consume this breakfast within 10 minutes. This meal has been designed to mimic the amount of energy (calories) and fat contained in a typical fast-food breakfast (e.g., from Tim Hortons or McDonalds). Each meal will provide 846 kcal, derived from 54 g fat (58% energy), 61 g carbohydrate (29% energy), and 29 g protein (13% energy).
  Interventions: Other: High-fat test meal

INTERVENTIONS:
Other: High-fat test meal — Ingestion of a mixed macronutrient breakfast meal providing 846 kcal, of which 58% is fat, 29% is carbohydrate and 13% is protein.

SUMMARY:
Long-term consumption (i.e., several weeks to months) of a diet that is high in fat (>35% daily calories from fat) is associated with the development of insulin resistance, a condition that can lead to a diagnosis of type 2 diabetes. Women tend to be better protected against the development of high-fat diet-induced insulin resistance compared with men, but it is not fully understand why this sex difference exists. It is possible that women metabolize high-fat meals differently than men, which might explain why they are less likely to develop type 2 diabetes over the course of their lifetime. However, no one has ever compared the metabolic response to a high-fat meal between men and women in the hours immediately after ingestion.

During this study, the investigators will administer a single high-fat "fast-food" style breakfast meal (846 kcal, of which 58% is fat) to 24 health young adults (n=12 men, n=12 women) 18-35 years old. Their objective is to determine whether there are differences in the way men and women metabolize high-fat meals, such as this one. The research team will take regular blood samples after participants ingest this meal to measure features of glucose metabolism (e.g., blood glucose and insulin) as well as resting oxygen uptake (VO2) measurements to examine how much of this meal is burned for energy in the hours immediately after ingestion.

DETAILED DESCRIPTION:
Long-term high-fat feeding is known to induce insulin resistance and impair whole-body glucose clearance in humans, yet knowledge of the glucose metabolic effects of high-fat feeding remains incomplete. Excess fat consumption leads to elevated circulating concentrations of non-esterified fatty acids (NEFAs), which (when taken up by muscle, an organ vital for glucose homeostasis) may interfere with insulin signaling and glucose disposal.

Despite the relatively rich body of research on high-fat feeding, the acute (i.e., 1-4 hours post-ingestion) effects of a high-fat meal on postprandial glucose metabolism are poorly characterized. Understanding the acute response to high-fat feeding is a key step towards uncovering the mechanisms that drive the development of dietary fat-induced insulin resistance. Limited work suggests that postprandial insulinemia may be elevated in response to a high-fat meal, and that this effect may be more pronounced in individuals with higher adiposity. Previous work has shown that ingestion of a mixed macronutrient meal high in saturated fat (~60% total fat, 32% saturated fat) stimulated significantly greater increases in circulating insulin concentrations in obese compared with lean middle-aged subjects. The effect of acute high-fat feeding on postprandial glycemia is less clear: studies have reported increased, decreased, or no change in glucose concentrations in response to a high-fat challenge. The quantity of fat administered may help explain these conflicting reports: studies have variously employed meals comprising 40%, 60% and up to 80% fat. These discrepancies in the literature may also be underpinned by the inclusion of males and females in the same study.

There is a paucity of data on the glucose metabolic response to high-fat feeding in human females. Although a handful of studies have included female subjects, this may have masked potentially divergent effects of high-fat feeding on glucose metabolism in males compared with females. Generally speaking, females have lower fasting plasma glucose concentrations (indicative of heightened hepatic insulin sensitivity) and are more adept at storing circulating NEFAs as subcutaneous adipose tissue (SAT). Although males have greater skeletal muscle mass (an important glucose reservoir) and lower whole-body adiposity than females, they preferentially accumulate adipose tissue in depots associated with metabolic dysfunction, such as the viscera and skeletal muscle [30]. Indeed, only one study to date has directly compared males and females to show that 7 days of suprarenergetic high-fat feeding (+50% kcal/d, 65% fat) stimulated an increase in trunk fat mass in males, with no discernable body composition changes in females. Given these sex-based differences in insulin sensitivity and adipose tissue storage, it is possible that females exhibit a distinct glucose metabolic response to high-fat feeding compared to males. However, this hypothesis has yet to be fully explored.

Therefore, in this study, the investigators will administer a single high-fat mixed macronutrient meal to a group of healthy young adults. Over the 4-hour postprandial period, they aim to compare the following in females versus males:

1. Circulating features of glucose metabolism (primary objective)
2. Circulating features of lipid metabolism (secondary objective)
3. Energy expenditure and substrate oxidation via indirect calorimetry (tertiary objective)

The investigators hypothesize that, compared with males, females will demonstrate:

1. Lower circulating concentrations of glucose, insulin, c-peptide and glucagon
2. Lower circulating concentrations of triglycerides, total cholesterol, low-density lipoprotein cholesterol and NEFAs; and higher circulating concentrations of high-density lipoprotein cholesterol
3. Greater energy expenditure and fat oxidation, and lower carbohydrate oxidation

This acute nutrition intervention study will involve a total of 3 visits to the laboratory (initial screening visit plus 2 study visits). After a screening visit to assess eligibility, young adults who have consented to participate will report to the laboratory after an overnight on 2 separate occasions: Baseline Assessment (Visit 1) and Nutrition Intervention (Visit 2).

Screening visit: Eligibility will be assessed during a screening session at the laboratory. The investigators will measure body mass, height, and resting blood pressure. Members of the research team will also help potential participants complete a Current Health Status Questionnaire, which will assess the potential participant's age, self-reported physical activity levels, and any medications or medical conditions that are relevant to the study.

Visit 1: Baseline Assessment: Participants will be asked to arrive after an overnight fast (i.e., no food or drink except for water for 8-12 hours). First, the investigators will perform a finger prick assessment to confirm eligibility and then evaluate body composition using dual-energy X-ray absorptiometry (DXA). Participants will be provided with a 3-day food diary and activity monitor at the conclusion of Visit 1, along with instructions on how to complete both.

Visit 2: Nutrition Intervention: After an overnight fast, participants will be asked to consume the high-fat test meal. The high-fat test meal will consist of bacon, eggs, cheese, tortilla, hashbrowns and mayonnaise (846 kcal, 58% fat, 29% carbohydrate, 13% protein). Members of the research team will prepare the meals in our metabolic kitchen. Before and after the meal is consumed, the researchers will take a series of blood samples and perform repeated resting VO2 measurements.

ELIGIBILITY:
Inclusion Criteria:

* BMI between 18.5 and 30.0 kg/m2
* Weight stable for the past 6 months (± 2kg)
* Exercise at or below the Canadian Physical Activity Guidelinesa
* Fasting blood glucose <6.0 mM
* Resting blood pressure <140/90 mmHg
* No hormone-altering contraceptive use (e.g., pill, patch, ring, injection)

Exclusion Criteria:

* Smoking
* Diabetes, cancer, or other metabolic disorders
* Cardiac or gastrointestinal problems
* Infectious disease
* Barium swallow or nuclear medicine scan in the previous 3 weeks
* Pregnant or breastfeeding
* Diagnosis of polycystic ovary syndrome
* Follow a vegan or vegetarian diet
* Not fully vaccinated against COVID19

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Estimated)
Dates: Start 2022-10-04 (Actual); Primary Completion 2027-05-30 (Estimated); Study Completion 2027-05-30 (Estimated)

PRIMARY OUTCOMES:
Plasma insulin | Will be measured in blood samples taken at 0 minutes (fasting), and 15, 30, 45, 60, 90, 120, 150, 180, 210, and 240 minutes post-ingestion of a high-fat meal
  Peak postprandial concentration and/or area under the curve
Plasma glucose | Will be measured in blood samples taken at 0 minutes (fasting), and 15, 30, 45, 60, 90, 120, 150, 180, 210, and 240 minutes post-ingestion of a high-fat meal
  Peak postprandial concentration and/or area under the curve
Plasma c-peptide | Will be measured in blood samples taken at 0 minutes (fasting), and 15, 30, 45, 60, 90, 120, 150, 180, 210, and 240 minutes post-ingestion of a high-fat meal
  Peak postprandial concentration and/or area under the curve
Plasma glucagon | Will be measured in blood samples taken at 0 minutes (fasting), and 15, 30, 45, 60, 90, 120, 150, 180, 210, and 240 minutes post-ingestion of a high-fat meal
  Peak postprandial concentration and/or area under the curve

SECONDARY OUTCOMES:
Plasma triglycerides | Will be measured in blood samples taken at 0 minutes (fasting), and 15, 30, 45, 60, 90, 120, 150, 180, 210, and 240 minutes post-ingestion of a high-fat meal
  Peak postprandial concentration and/or area under the curve
Plasma cholesterols (total and HDL) | Will be measured in blood samples taken at 0 minutes (fasting), and 15, 30, 45, 60, 90, 120, 150, 180, 210, and 240 minutes post-ingestion of a high-fat meal
  Peak postprandial concentration and/or area under the curve
Plasma non-esterified fatty acids | Will be measured in blood samples taken at 0 minutes (fasting), and 15, 30, 45, 60, 90, 120, 150, 180, 210, and 240 minutes post-ingestion of a high-fat meal
  Peak postprandial concentration and/or area under the curve
Respiratory exchange ratio (RER) | Will be measured using indirect calorimetry and a facemask at -10 to 0 minutes (fasting), and 50-60 minutes, 110-120 minutes, 170-180 minutes and 230-240 minutes post-ingestion of a high-fat meal.
  Average resting RER over a 10-minute sampling period

CONTACTS AND LOCATIONS:
Overall Officials: Kirsten E Bell, PhD, Principal Investigator — McMaster University
Locations (1):
- McMaster University, Hamilton, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No
No IPD will be shared with anyone outside of the research team.

REFERENCES:
- [Background] Whytock KL, Parry SA, Turner MC, Woods RM, James LJ, Ferguson RA, Stahlman M, Boren J, Strauss JA, Cocks M, Wagenmakers AJM, Hulston CJ, Shepherd SO. A 7-day high-fat, high-calorie diet induces fibre-specific increases in intramuscular triglyceride and perilipin protein expression in human skeletal muscle. J Physiol. 2020 Mar;598(6):1151-1167. doi: 10.1113/JP279129. Epub 2020 Feb 14. PMID 31958145
- [Background] Bachmann OP, Dahl DB, Brechtel K, Machann J, Haap M, Maier T, Loviscach M, Stumvoll M, Claussen CD, Schick F, Haring HU, Jacob S. Effects of intravenous and dietary lipid challenge on intramyocellular lipid content and the relation with insulin sensitivity in humans. Diabetes. 2001 Nov;50(11):2579-84. doi: 10.2337/diabetes.50.11.2579. PMID 11679437
- [Background] Lundsgaard AM, Fritzen AM, Sjoberg KA, Kleinert M, Richter EA, Kiens B. Small Amounts of Dietary Medium-Chain Fatty Acids Protect Against Insulin Resistance During Caloric Excess in Humans. Diabetes. 2021 Jan;70(1):91-98. doi: 10.2337/db20-0582. Epub 2020 Oct 29. PMID 33122393
- [Background] Chiu CH, Yang TJ, Chen CH, Zeng MJ. High fat meals increases postprandial fat oxidation rate but not postprandial lipemia. Lipids Health Dis. 2019 Oct 23;18(1):182. doi: 10.1186/s12944-019-1129-x. PMID 31647036
- [Background] Ando T, Nakae S, Usui C, Yoshimura E, Nishi N, Takimoto H, Tanaka S. Effect of diurnal variations in the carbohydrate and fat composition of meals on postprandial glycemic response in healthy adults: a novel insight for the second-meal phenomenon. Am J Clin Nutr. 2018 Aug 1;108(2):332-342. doi: 10.1093/ajcn/nqy086. PMID 29924301
- [Background] Parry SA, Turner MC, Woods RM, James LJ, Ferguson RA, Cocks M, Whytock KL, Strauss JA, Shepherd SO, Wagenmakers AJM, van Hall G, Hulston CJ. High-Fat Overfeeding Impairs Peripheral Glucose Metabolism and Muscle Microvascular eNOS Ser1177 Phosphorylation. J Clin Endocrinol Metab. 2020 Jan 1;105(1):dgz018. doi: 10.1210/clinem/dgz018. PMID 31513265
- [Background] Whytock KL, Shepherd SO, Cocks M, Wagenmakers AJM, Strauss JA. Young, healthy males and females present cardiometabolic protection against the detrimental effects of a 7-day high-fat high-calorie diet. Eur J Nutr. 2021 Apr;60(3):1605-1617. doi: 10.1007/s00394-020-02357-3. Epub 2020 Aug 13. PMID 32789769
- [Background] Alayón, A. N. et al. Impacto metabólico e inflamatorio de una comida rica en grasas saturadas y su relación con la obesidad abdominal. Biomédica 38, 100-107, doi:10.7705/biomedica.v38i0.3911 (2017).
- [Background] Wang F, Lu H, Liu F, Cai H, Xia H, Guo F, Xie Y, Huang G, Miao M, Shu G, Sun G. Consumption of a liquid high-fat meal increases triglycerides but decreases high-density lipoprotein cholesterol in abdominally obese subjects with high postprandial insulin resistance. Nutr Res. 2017 Jul;43:82-88. doi: 10.1016/j.nutres.2017.05.010. Epub 2017 May 17. PMID 28673468
- [Background] Obeid R, Awwad HM, Knell AI, Hubner U, Geisel J. Glucose and Fat Tolerance Tests Induce Differential Responses in Plasma Choline Metabolites in Healthy Subjects. Nutrients. 2018 Sep 1;10(9):1209. doi: 10.3390/nu10091209. PMID 30200465